CLINICAL TRIAL: NCT01593553
Title: Systematic ECG Screening for Atrial Fibrillation Among 75 Year Old Subjects in the Region of Stockholm and Halland, Sweden.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Professor Mårten Rosenqvist, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Strokestop
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Screening; Stroke prevention; Cost effectiveness
MeSH Terms: conditions — Atrial Fibrillation; Stroke

ARMS (2):
- ECG screening (Experimental): Twice daily screening using intermittent ECG recorder (Zenicor) for two weeks
  Interventions: Other: ECG screening for atrial fibrillation using intermittent ECG recorder
- Control group (No Intervention): Standard of care

INTERVENTIONS:
Other: ECG screening for atrial fibrillation using intermittent ECG recorder — ECG screening for atrial fibrillation with intermittent ECG recording (Zenicor device) for 14 days. Introduction of anticoagulants in the case of atrial fibrillation.
  Other Names: Zenicor ECG recorder
  Arms: ECG screening

SUMMARY:
The purpose of this study is to determine whether screening for atrial fibrillation by intermittent ECG recording and initiation of anticoagulation treatment among high risk individuals is cost-effective and can lower the incidence of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 75-76 years of age living in the region of Stockholm or Halland

Exclusion Criteria:

* Not fulfilling the inclusion criteria

Ages: 75 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7173 (Actual)
Dates: Start 2012-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Ischaemic or haemorrhagic stroke, systemic embolism, major bleeding leading to hospitalization or death from any cause | Five years. Interim analysis after 3 years.
  A composite endpoint of incidence of ischamemic and haemorrhagic stroke, incidence of systemic embolism, major bleeding requiring hospitalization and all cause mortality in the group randomized to screening compared to the control group

SECONDARY OUTCOMES:
Ischaemic stroke | Five years. Interim analysis after 3 years.
  Incidence of ischaemic stroke in the group randomized to screening compared to the control group
Ischaemic stroke and systemic thromboembolism | Five years. Interim analysis after 3 years.
  Incidence of ischaemic stroke and systemic thromboembolism in the group randomized to screening compared to the control group
Ischaemic stroke and systemic thromboembolism | Five years. Interim analysis after 3 years.
  Incidence of ischaemic stroke and systemic thromboembolism in the group participating in screening (as treated) compared to the control group
Dementia | Five years. Interim analysis after 3 years.
  Incidence of dementia in the group randomized to screening compared to the control group
All cause mortality | Five years. Interim analysis after 3 years.
  All cause mortality in the group randomized to screening compared to the control group
Cardiovascular mortality | Five years. Interim analysis after 3 years.
  Cardiovascular in the group randomized to screening compared to the control group
Hospitalization due to cardiovascular disease | Five years. Interim analysis after 3 years.
  Hospitalization due to cardiovascular disease in the group randomized to screening compared to the control group
Ischaemic or haemorrhagic stroke, systemic embolism, major bleeding leading to hospitalization, hospitalization due to cardiovascular disease or death from any cause | Five years. Interim analysis after 3 years.
  In the group randomized to screening compared to the control group
Cost effectivity | Five years
Initiation and compliance to oral anticoagulation therapy | Five years
  The National Prescription Drug's register will be used to study intiation and duration of oral anticoagulation therapy in a as-treated and per-protocol analysis in the screened population compared to the control group
Detection of atrial fibrillation | Five years
  Incidence of atrial fibrillation in the group randomized to screening compared to the control group
Pulmonary embolism and deep vein thrombosis | Five years
  Incidence of pulmonary embolism and deep vein thrombosis in the group randomized to screening compared to the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Trial Alliance, KTA Prim, Stockholm, Sweden

REFERENCES:
- [Derived] Svennberg E, Friberg L, Frykman V, Al-Khalili F, Engdahl J, Rosenqvist M. Clinical outcomes in systematic screening for atrial fibrillation (STROKESTOP): a multicentre, parallel group, unmasked, randomised controlled trial. Lancet. 2021 Oct 23;398(10310):1498-1506. doi: 10.1016/S0140-6736(21)01637-8. Epub 2021 Aug 29. PMID 34469764
- [Derived] Hygrell T, Stridh M, Friberg L, Svennberg E. Prognostic Implications of Supraventricular Arrhythmias. Am J Cardiol. 2021 Jul 15;151:57-63. doi: 10.1016/j.amjcard.2021.04.020. PMID 34167689
- [Derived] Svennberg E, Henriksson P, Engdahl J, Hijazi Z, Al-Khalili F, Friberg L, Frykman V. N-terminal pro B-type natriuretic peptide in systematic screening for atrial fibrillation. Heart. 2017 Aug;103(16):1271-1277. doi: 10.1136/heartjnl-2016-310236. Epub 2017 Mar 2. PMID 28255099
- [Derived] Svennberg E, Engdahl J, Al-Khalili F, Friberg L, Frykman V, Rosenqvist M. Mass Screening for Untreated Atrial Fibrillation: The STROKESTOP Study. Circulation. 2015 Jun 23;131(25):2176-84. doi: 10.1161/CIRCULATIONAHA.114.014343. Epub 2015 Apr 24. PMID 25910800